CLINICAL TRIAL: NCT00519246
Title: Clinical Comparison of Postoperative Pain Therapeutic Effects After Benign Mastectomy
Brief Title: Comparison of Pain Therapeutic Effects After Benign Mastectomy
Acronym: COPTEAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Maternal and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-2579-4FW; NMCH2007-241
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Pain, Postoperative; Mastectomy
Keywords: Breast Neoplasms; Non-Steroidal Anti-Inflammatory Agents; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms; Agnosia | interventions — Sodium Chloride; Analgesics, Opioid; Anti-Inflammatory Agents, Non-Steroidal; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- I (Placebo Comparator): No drug was delivered.
  Interventions: Drug: Saline
- II (Active Comparator): Butorphanol tartrate 1mg was given intravenously.
  Interventions: Drug: Opioid
- III (Active Comparator): Butorphanol tartrate 2 mg was given intravenously.
  Interventions: Drug: Opioid
- IV (Active Comparator): Flurbiprofen Axetil 50 mg was given intravenously.
  Interventions: Drug: NSAID
- V (Active Comparator): Flurbiprofen Axetil 100 mg was given intravenously.
  Interventions: Drug: NSAID
- VI (Active Comparator): Tramadol Hydrochloride 10 mg was given intravenously.
  Interventions: Drug: Opioid
- VII (Active Comparator): Tramadol Hydrochloride 20 mg was given intravenously.
  Interventions: Drug: Opioid

INTERVENTIONS:
Drug: Saline — Saline 5 ml administrated intravenously
  Other Names: Physiological solution
  Arms: I
Drug: Opioid — Butorphanol tartrate 1 mg i.v.
  Other Names: NuoYang
  Arms: II
Drug: Opioid — Butorphanol Tartrate 2 mg i.v.
  Other Names: NuoYang
  Arms: III
Drug: NSAID — Flurbiprofen Axetil 50 mg i.v.
  Other Names: CaiFen
  Arms: IV
Drug: NSAID — Flurbiprofen Axetil 100 mg i.v.
  Other Names: CaiFen
  Arms: V
Drug: Opioid — Tramadol Hydrochloride 10 mg i.v.
  Other Names: Trama
  Arms: VI
Drug: Opioid — Tramadol Hydrochloride 20 mg i.v.
  Other Names: Trama
  Arms: VII

SUMMARY:
With the incremental trend of benign breast tumor, the surgical process of mastectomy was proceeded too much every day, especially in the Maternal Health Care Hospital, but whether the investigators can find another way to relieve the postoperative pain after such an operation is still unknown. The investigators hypothesized that the pain from the relatively small surgery may not be significant compared to different treatments, even if no drug was delivered to them. The investigators are enrolling patients who underwent mastectomy from benign breast tumor, and are observing the analgesic effects of different drugs.

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* No cardiac and pulmonary diseases
* ASA I-II
* No alcohol drinking.

Exclusion Criteria:

* <19yrs, and >65yrs
* History of central active drugs administration
* Drug abuse
* Hypertension
* Diabetes
* Any other chronic diseases.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2000 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) rating of pain | 0-24h after surgeries

SECONDARY OUTCOMES:
VAS rating of sedation | 0h to 24h after the end of the operation
Overall VAS rating of satisfaction with analgesia | 24 h after operation
Incidence of side effects | From the initiation of analgesia (0 h) to the end of the study (24 h postoperative)

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Care Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Shen X, Wang F, Xu S, Ma L, Liu Y, Feng S, Wang W, Zhao Q, Li X, Zhao L, Yao X, Qu J, Xie B, Wang H, Yuan H, Cao Y, Sun Y, Wang W, Guo L, Song Z, Wang Z, Guan X. Comparison of the analgesic efficacy of preemptive and preventive tramadol after lumpectomy. Pharmacol Rep. 2008 May-Jun;60(3):415-21. PMID 18622068